CLINICAL TRIAL: NCT05958953
Title: PeRinatal Outcomes With ACTive Versus Expectant Management of Women With Pre-labor Rupture Of Membranes: a Phase III, Open-label, Randomized Controlled Multicentric Trial
Brief Title: PeRinatal Outcomes With ACTive Versus Expectant Management of Women With Pre-labor Rupture Of Membranes
Acronym: PROACT PROM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Prof. Fabio Facchinetti, Full professor of Obstetrics and Gynecology Chairmen Unit of Obstetrics and Gynecology, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-002480-30
Record Dates: First submitted 2023-06-06; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Rupture of Membranes; Premature; Distress; Fetal, Complicating Delivery; Delayed Delivery After Spontaneous or Unspecified Rupture of Membranes; Maternal Sepsis
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Pregnancy Complications, Infectious | interventions — Labor, Induced

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active management (Experimental): early IOL within 8 hours of rupture of membranes. Center-specific IOL protocols will be used.
  Interventions: Procedure: Induction of Labor IoL
- Expectant management (No Intervention): monitoring until 24 hours from rupture of membranes, with subsequent induction of labor (IOL).

INTERVENTIONS:
Procedure: Induction of Labor IoL — Center-specific IOL protocols, based on international guidelines, will be used.
  Arms: active management

SUMMARY:
Term pre-labor rupture of membranes (PROM) occurs in about 12% of pregnancies and the time between PROM and delivery increases the risk of maternal/fetal infections. However, conflicting results are reported by studies investigating risks and benefits of expectant management versus induction of labor (IOL). Expectant management was associated with maternal and fetal infectious complications and subsequent increased risk of maternal and neonatal morbidity. Studies suggest that the increase in infectious risk for both is proportional to the increase in the time interval between the ROM and the birth, others reject this assumption.

In PeRinatal Outcomes With ACTive Versus Expectant Management of Women With Pre-labor Rupture Of Membranes (PROACTIVE PROM) on admission, PROM will be diagnosed. After 6 hours from the rupture of membranes, the woman will then be assessed for eligibility. A 1:1 randomization will follow within two hours (6-8 hours from PROM) in two distinct arms: 1) Expectant management 2) Active menagement (early IOL within 8 hours of rupture of membranes).

The first objective of this study is to evaluate whether active management of women with PROM (early induction) reduces the newborn need of respiratory support.

The secondary objectives of this study are related to the safety of the active management assessed through the rate of stillbirths, the onset of infections in both mother and fetus and the length of hospitalization of the dyads. Moreover, another objective is to reduce the use of antibiotic treatments (ATB) in both mothers and newborns.

The rationale of this study is that reducing the time between the PROM and delivery through an early IOL will reduce the adverse maternal and neonatal outcomes.

The hypothesis underneath this trial comes from a preliminary retrospective cohort study conducted in Modena, which included 2689 mother-neonates dyads from singleton pregnant women at term. In deliveries of ROM >24 hours significantly more neonates required ventilatory support than those born within 24 hours, although no significant differences were found regarding overt infections. According to the Cochrane database, expectant management of PROM is associated with maternal and fetal infectious complications and subsequent increased risk of maternal and neonatal morbidity together with an increased risk of ATB use. The increase of infectious risk is proportional to the time elapsed since the rupture of the membranes (ROM) and birth. However, unpublished data from our group suggest that respiratory distress requiring interventions may be frequently caused by intrinsic inflammatory-related effects of prolonged ROM rather than infection; this is suggested by an increase of C-reactive protein levels in neonates with mild respiratory signs untreated with antibiotics.

In addition, in a survey performed in our country expectant management increased intrapartum antibiotic prophylaxis (IAP), although not strictly indicated by the most current guidelines.

On the light of these data, it appears reasonable to promote induction of labor, to prevent complication caused not only by the infectious risk mentioned above, but also respiratory distress, probably associated to a neonatal maladaptation, in non-infectious newborns.

On the other hand, it should also be considered that 75% of women enter labor spontaneously within 24 hours from PROM and induction of labor (IOL) might not be needed in such cases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age at the time of randomization
2. Gestational age ≥ 37 weeks
3. Negative rectovaginal GBS swab
4. Absent/poor uterine contractile activity 6 h after PROM (0-2 contractions /10 min)
5. Cephalic presentation
6. Ability to provide an informed consent
7. Signed informed consent

Exclusion Criteria:

1. Prematurity (<37 weeks)
2. GBS positive vagino-rectal swab or with an unknown swab
3. Multiple pregnancies
4. Previous cesarean section (CS)
5. Breech presentation, transverse lie or other indication for elective CS
6. Suspected clinic for intra-amniotic infection (According to the Triple I criteria)
7. Stained amniotic fluid
8. Alterations of the FHR
9. Unknown exact ROM time
10. Known hypersensitivity to drugs for IOL or their excipients
11. Presence of unknown vaginal bleeding
12. Presence of maternal kidney disease (GFR <15 ml/min/1,73 m2).
13. Every condition contraindicating vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
Rate of respiratory support in newborns | On day 1 or 2 post-partum all relevant delivery and post-partum as well as neonatal variables will be collected.
  The primary objective of this study is to evaluate whether active management of women with PROM (early induction) reduces the newborn need of respiratory support, collecting data on Apgar score, neonatal blood gas analysis and the rate of respiratory distress after birth and rate of respiratory support divided by type. The need for neonatal ventilatory support will be evaluated at delivery and include at least one of the following measures: free flowing oxygen in incubator, low flow oxygen (<2 LPM), high flow oxygen (>3 LPM), NCPAP or other NIV, mechanical ventilation.

SECONDARY OUTCOMES:
Stillbirth and infection rate | On day 1 or 2 post-partum all relevant delivery and post-partum as well as neonatal variables will be collected.
  This secondary objectives of this study are related to the safety of the active management assessed through the rate of stillbirths, the onset of infections in the mother and fetus and through the length of hospitalization of the dyads. Moreover, another objective is to reduce the use of antibiotic treatments (ATB) in both mothers and newborns.
length of hospitalization expressed in days | From day 1 after delivery to the end of the puerperium (42 days after delivery)
  The lenght of hospitalization and the need for re-hospitalizations are related to the safety of the active management assessed through the rate of stillbirths, the onset of infections in the mother and fetus and through the length of hospitalization of the dyads. Moreover, another objective is to reduce the use of antibiotic treatments (ATB) in both mothers and newborns.
use of antibiotics in both mother and newborn as quantity (mg) and quality. | From admission in the Hospital to 42 days after delivery
  The use of antibiotics will be recorded
neonatal infection as the yield of pathogen from blood or CFS coltures | From birth to 42 days after delivery
  Suspected infection is based on the presence of clinical symptoms (neonatal tachycardia, hyperpyrexia, alteration of the skin color) and abnormal laboratory markers, i.e. an increase in C reactive proteins above 1.5 mg/dl.
Rate of Pathogen isolation in placenta's speciemen | Collection of speciemens immediately after delivery
  Placentas and umbilical cord will be collected only in the Milano Buzzi center

CONTACTS AND LOCATIONS:
Locations (1):
- AUO Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided